CLINICAL TRIAL: NCT05265286
Title: A Phase II, Multicentre, Open-label Study to Evaluate the Pharmacokinetic, Safety and Preliminary Efficacy of PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection in Subjects With Severe Hemophilia A
Brief Title: A Study of Repeat Dosing of PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Gensciences lnc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTR20220283
Record Dates: First submitted 2022-02-22; First posted 2022-03-03 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Severe Hemophilia A
Keywords: Pharmacokinetics;; Safety;; immunogenicity;; Preliminary efficacy
MeSH Terms: conditions — Hemophilia A | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 prophylaxis treatment (Experimental): Subjects of high dose group are being received four doses of FRSW117. dosing on day1(ED1), day8(ED2), day15(ED3), day22(ED4) respectively.
  Subjects of low dose group are being received four doses of FRSW117. dosing on day1(ED1), day8(ED2), day15(ED3), day22(ED4) respectively.
  All subjects are being received PK assessment in ED1 and ED4.
  Interventions: Drug: FRSW117

INTERVENTIONS:
Drug: FRSW117 — Subjects of high dose group are being received four doses(50 IU/kg,once a week or every 7 days) of FRSW117.
  Subjects of low dose group (40 IU/kg,once a week or every 7 days)are being received four doses of FRSW117.
  Other Names: PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection

SUMMARY:
Primary objective: To assess the pharmacokinetics, Safety and immunogenicity of Repeat Dosing of PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection With Severe Hemophilia A(FRSW117) Secondary objectives: To assess Preliminary efficacy of Repeat Dosing of PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for Injection With Severe Hemophilia A.

ELIGIBILITY:
Key Inclusion Criteria:

* The activity of the coagulation factor VIII (FVIII:C) < 1%.
* Patients previously treated with FVIII concentrate (s) for a minimum of 150 exposure days (EDs) prior to study entry
* Normal prothrombin time or INR < 1.3
* Negative lupus anticoagulant

Key Exclusion Criteria:

* Hypersensitive to any of the excipients of the test materials (e.g. allergic to murine or hamster origin heterologous proteins)
* History of hypersensitivity or anaphylaxis associated with any FVIII or II immunoglobulin administration
* Current FVIII inhibitor-positive or history of FVIII inhibitor-positive
* Other coagulation disorder(s) in addition to hemophilia A.• Significant hepatic or renal impairment (ALT and AST > 2×ULN; serum bilirubin level > 2 × upper limit of normal (ULN), Urea /BUN > 2×ULN, Cr > 176.8 µmol/L)
* One or more clinically significant tests for Human Immunodeficiency Virus (HIV), Antisyphilitic spirulina (TPHA) and Hepatitis C Virus (HCV) Antibody
* Patients who received any anticoagulant or antiplatelet therapy within one week prior screening or need to receive an anticoagulant or antiplatelet therapy during the period of clinical trials
* Patients having major surgery or receiving blood or bood components transfusion within 4 weeks prior screening or having planned major surgery schedule during the study
* Patients who previously participated in the other clinical trials within one month prior screening
* Any life-threatening disease or condition which, according to the investigator's judgment, could not benefit from the trial participation
* Patient who is considered by the other investigators not suitable for clinical study

Other protocol-defined inclusion/exclusion Criteria May Apply.

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Hemophilia A is an X-chromosome-linked recessive inherited bleeding disorder caused by a deficiency of coagulation factor VIII (FVIII)
Enrollment: 15 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2022-08-21 (Actual); Study Completion 2022-08-21 (Actual)

PRIMARY OUTCOMES:
Maximum measured concentration of FVIII:C (Cmax) | Pre-dose and post dose up to 10 days
  Measured by One-Stage Clotting Assay
Time required for the concentration of the drug to reach half of its original value (T1/2) | Pre-dose and post dose up to 10 days
  Measured by One-Stage Clotting Assay
Area Under the Curve to Infinity (AUC) | Pre-dose and post dose up to 10 days
  Measured by One-Stage Clotting Assay
The measure of the efficiency of the body to remove the drug and the unit is the volume of the plasma or blood cleared of drug per unit time (CL) | Pre-dose and post dose up to 10 days
  Measured by One-Stage Clotting Assay
Evaluation of the level of anti-PEG-rFⅧFc antibody production in participants | Pre-dose and post dose up to 36 days
Evaluation of the level of anti-PEG antibody production in participants | Pre-dose and post dose up to 36 days

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE V5.0 | Pre-dose and post dose up to 36 days
  Adverse events related to PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein according to Common Terminology Criteria for Adverse Events (CTCAE) NCI.V5.0.
Development of Inhibitor | Pre-dose and post dose up to 36 days
  Measured by the Nijmegen-Modified Bethesda Assay
score of bleeding symptoms and Vital signs | Pre-dose and post dose up to 36 days
  Response to treatment with PEG Recombinant Human Coagulation Factor VIII-Fc Fusion Protein for bleeding episodes, using the 4-point bleeding response scale

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, PhD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College.
Locations (5):
- China (5):
  - People'S Hospital of Zhengzhou, Zhengzhou, Henan
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - People'S Hospital of Rizhao, Rizhao, Shandong
  - Institute of Hematology & Blood Diseases Hospital Chinese Academy of Medical Sciences & Peking Union Medical College., Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No